CLINICAL TRIAL: NCT02101307
Title: A Multi-center Non-interventional Study in Rheumatoid Arthritis (RA) Patients Treated With Tocilizumab
Brief Title: Multicenter, Post-marketing, Non-interventional, Observational Study in RA Patients Treated With RoActemra/Actemra (Tocilizumab)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28429
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- RA Patients on RoActemra/Actemra treatment

SUMMARY:
This non-interventional study will observe the usage and efficacy of RoActemra/Actemra in patients with rheumatoid arthritis (RA) who have recently begun treatment. The treatment regimen will be directed by the treating physician according to clinical practice. Patients are expected to be observed for approximately 6 months after beginning treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age
* Patients with a diagnosis of moderate to severe RA according to the revised (1987) ACR criteria
* Patient in whom the treating physician has made the decision to commence RoActemra/Actemra treatment (in accordance with the local label). This can include patients who have received RoActemra/Actemra treatment within 8 weeks prior to the enrolment visit
* Patient has given informed consent

Exclusion Criteria:

* Patients who have received RoActemra/Actemra more than 8 weeks prior to the enrolment visit
* Patients who have previously received RoActemra/Actemra in a clinical trial or for compassionate use
* Patients who have received treatment with any investigational agent within 4 weeks (or 5 half-lives of investigational agent, whichever is longer) before starting treatment with RoActemra/Actemra
* Patients with a history of autoimmune disease or of any joint inflammatory disease other than RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with rheumatoid arthritis starting RoActemra/Actemra treatment
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-07-09 (Actual); Primary Completion 2017-05-22 (Actual); Study Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
Proportion of patients on RoActemra/Actemra treatment 6 months after treatment initiation | 6 months

SECONDARY OUTCOMES:
Proportion of patients with systemic manifestation of RA | At Baseline
Record of RA treatment history | 6 months
Treatment patterns during observation period, assessed by alteration in dosing regimen | 6 months
Efficacy as assessed by total joint count evaluation | 6 months
Incidence of adverse events | 6 months
Health-related quality of life as assessed by questionnaire | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- China (25):
  - Peking University First Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Union Hospital, Beijing
  - Xiangya Hospital of Centre-South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - Sichuan Provincial People's Hospital, Chengdu
  - Southwest Hospital , Third Military Medical University, Chongqing
  - Sun Yat-sen Memorial Hospital, Guangzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - The First Affiliated Hospital of Jinan University, Guangzhou
  - TCM-Integrated Hospital of Southern Medical University, Guangzhou
  - Zhejiang People's Hospital, Hangzhou
  - Affiliated Hospital of Inner Mongolia Medical College, Hohhot
  - The First People's Hospital of Yunnan Province, Kunming
  - The First Affiliated Hospital of Henan UN of Science and Technology, Luoyang
  - Affiliated Hospital of North Sichuan Medical College, Nanchong
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Futian District people's Hospital of Shenzhen City, Shenzhen
  - Xinjiang Uygur Autonomous Region People Hospital, Ürümqi
  - Tongji Hosp, Tongji Med. Col, Huazhong Univ. of Sci. & Tech, Wuhan
  - Wuxi People's Hospital, Wuxi
  - The Second Affiliated Hospital of The Fourth Military Medical University (Tangdu Hospital), Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - YanTaishan Hospital of Yantai City, Yantai
  - Zhuzhou Central Hospital, Zhuzhou